CLINICAL TRIAL: NCT03586206
Title: Relationship Between C. Difficile Toxins' Serum Level With C. Difficile Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Roma Tre University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MISP57289
Record Dates: First submitted 2018-05-28; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-05

CONDITIONS: Clostridium Difficile; Clostridium Difficile Infection
Keywords: Clostridium difficile; toxins; serum; infection
MeSH Terms: conditions — Clostridium Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild-moderate C.difficile infection
- severe C.difficile infection
- severe complicated/fulminant C.difficile infection

SUMMARY:
To assess the association between Clostridium difficile (CD) toxins' serum levels and the grade of Clostridium difficile infection (CDI) severity/failure to CDI treatment and rate of recurrence. Furthermore, the kinetics of CD toxins in serum of CDI patients undergoing anti-CDI treatment, as well as the relationship between serum toxins levels and length of CDI diarrhea will be evaluated.

DETAILED DESCRIPTION:
Background. C. difficile frequently induces toxemia, however due to limited sensitivity of existing diagnostic tools, it goes undetected in common clinical practice. Although undetected, Clostridium difficile infection (CDI)-induced toxemia is often experienced, and this explains the systemic complications of life-threatening CDI cases. Until recently, although the pathogenetic process was already known, the phenomenon of extraintestinal damage caused by C. difficile toxins has been undervalued. However, a recent study has proven toxemia in humans. In the last 5 years, animal studies have proven the presence of C. difficile toxins in several body fluids, toxemia correlating with systemic disease and mortality. However, although toxin A (TcdA) and B (TcdB) are the primary virulence factors responsible for C. difficile-associated diarrhea and inflammation, only three toxemia-positive cases (two adults and one child) have been reported so far in humans. The explanation for such a low number of toxemia-positive cases may be the lack of sensitive toxins detection method.

Objectives.

1. To assess the association between CD toxins' serum levels and grade of CDI severity/failure to CDI treatment and rate of recurrence.
2. To evaluate the kinetics of CD toxins in serum of CDI patients undergoing anti-CDI treatment.
3. To assess the relationship between serum toxins levels and length of CDI diarrhoea.

Study design. Prospective observational study on the measurement of serum levels of CD toxins in patients with CDI.

In order to assess the relationship between C difficile toxins' serum level and severity and recurrence rate, 45 consecutive patients with documented CDI infection will be studied, including 20 with mild-moderate CDI, 20 with severe CDI, and 5 with severe complicated/fulminant CDI according to ESCMID definition. For each patient three determination of serum toxins will be performed at time 0 (before initiation of anti-CDI treatment), 4d, 10d.

Patients will be followed up to three months after the recovery from the first episode.

The serum toxins' levels will be correlated to severity and to the first recurrence.

Methodology

1. Serum samples Peripheral blood will be obtained from each healthy and CDI subjects. Serum will be separated from the peripheral blood sample by centrifugation at 700 g for 5 min, and then stored at -20°C until measurement.
2. Serum IgG depletion It has been reported that neutralizing antibodies present in human serum, mostly IgG, are able to mask the C. difficile toxins levels in serum. Total IgG in serum samples will be removed with Protein A beads (Santa Cruz Biotechnology, Santa Cruz, CA, USA). Two milliliters of human serum sample will be applied to an equal volume of protein A beads resuspended in binding buffer, and incubated at room temperature under rotary agitation for 1 h. The IgG bound to the Protein A beads will be removed by centrifugation. The proper IgG depletion will be evaluated by western blot.
3. SDS-PAGE and western blot IgG-purified sera will be resolved by 10% SDS-PAGE and transferred onto PVDF membranes (Bio-Rad, Hercules, CA, USA). After blocking for 1 h at room temperature (RT) with 5% non-fat dry milk (w/v) and 0.5% Tween-20 (v/v) dissolved in PBS, membranes will be probed with anti-human IgG primary antibody (anti-Human IgG, γ-chain specific antibody; Sigma-Aldrich, St. Louis, MO, USA), at 4°C overnight. Membranes will be then incubated for 1 h at RT with the HRP-conjugated secondary antibody (Bio-Rad). Proteins will be visualized by the enhanced chemiluminescence (ECL) detection system (Bio-Rad) and images will be acquired using the Chemidoc System (Bio-Rad).
4. Dot-blot

d1. Standard reference The dot-blot condition set-up for the evaluation of C. difficile TcdA and TcdB levels in the human serum samples will be performed as follows. Recombinant TcdA and TcdB (Enzo Life Science, Farmingdale, NY) will be dissolved in deionized water to obtain 0.2 mg/mL stock solutions. Toxins will be serially diluted from 0.001 pg to 1000 pg in PBS at pH 7.4. Ten microliters of diluted TcdA and TcdB will be blotted in triplicate into EMD Millipore MultiScreen™ 96-Well Assay Plates (Fisher Scientific, Waltham, MA, USA). After 10 min of drying, the membrane will be immersed in 2% BSA-PBS (w/v) buffer for 1 h at 37 °C. The membrane will be washed with PBS containing 0.05% Tween 20, at pH 7.2) for 2 min and immersed in anti-C. difficile TcdA and anti-C.difficile TcdB (Abcam) primary antibodies (recognizing the native proteins), for 1 h at RT. The proper dilution of the anti-TcdA and -TcdB antibodies will be tested, according to manufacturer's instructions. The membrane will be then washed for 2 min and the dots corresponding to the increasing concentrations of TcdA and TcdB will be visualized by ECL and acquired by the Chemidoc system. The intensities of the colored blots will be considered as a standard reference to evaluate the minimum concentration of TcdA and TcdB that can be detected by this method.

d2. Set-up of the volume and dilution of human serum to be used The sensitivity of the method will be assessed using toxemia-negative spiked human serum samples freshly prepared by adding recombinant toxins (positive control). The quantity of recombinant TcdA and TcdB to be added to the spiked serum will be chosen on the basis of results obtained in the previous section (d1). This will allow determining: (i) the minimal concentration of TcdA and TcdB that can be detected by the dot-blot method when diluted in the human serum; and (ii) the proper volume and dilution of the human serum to be added to each well of the MultiScreen™ 96-well assay plates.

d3. Dot blot on the serum samples of CDI patients to determine toxins levels Human sera derived from CDI patients will be IgG-depleted (see section b) and then spotted trice into the MultiScreen™ 96-well assay plates. The dot-blot method described in section d1 will be applied to determine and semi-quantify TcdA and TcdB levels, using the TcdA and TcdB standard curves.

ELIGIBILITY:
Inclusion Criteria:

* 45 consecutive patients with documented CDI infection, including:
* 20 with mild-moderate CDI
* 20 with severe CDI
* 5 with severe complicated/fulminant CDI, according to ESCMID definition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2019-09-15 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Setup of the method. | For each patient, the change of serum toxins levels after 4 and 10 days from the initation of anti-CDI treatment will be compared to levels before initation of anti-CDI treatment.
  Mann-Whitney U-tests will be used to compare the intensity of each triplicate chemiluminescent spot of the CDI serum tested with the TcdA and TcdB standard curves, and to compare the intensities of the chemiluminescent spots of CDI patients with those of normal subjects. Quantitative variables will be expressed as the median and IQR.
Validation on the proposed method | The proposed method will be compared with reference tests evaluating change of serum toxins levels after 4 and 10 days from the initiation of anti-CDI treatment with levels before initiation of anti-CDI treatment.
  According to ESCMID guidelines, our method will be compared with reference tests that are defined as the best tests currently available for CDI diagnosis (i.e., cell cytotoxicity neutralization assay (CCNA) and toxigenic culture (TC)). As both these reference tests detect different things, and because of this they will not necessarily agree with each other in all samples, results for each reference test will be analysed separately.
Performance of the proposed method | The evaluation of the performance of the proposed method will be assed by evaluating the change of toxins levels from baseline levels (time 0) at 4 and 10 days from the initiation of anti-CDI treatment.
  The performance of our method will be assessed using the receiver operating characteristic (ROC) curve and the area under the curve (AUC). The sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of the prediction rule of poor outcome will be calculated. Validity values will be calculated with a 95% CI following an exact binomial distribution. A P value <0.05 will be considered significant
Correlation of toxins kinetics and CDI severity | Determination of serum toxin kinetics will be evaluated by the change from baseline levels (time 0) at 4 and 10 days from the initiation of anti-CDI treatment. For recurrence rate, the follow up will be of 30 days after cessation of diarrhea.
  Toxin kinetics (TcdA alone, TcdB alone, TcdA+TcdB) will be correlated by one-way analysis of variance (ANOVA) with CDI severity (defined according to ESCMID guidelines)
Correlation between toxins levels and the duration of diarrhea | Determination of serum toxin kinetics will be evaluated by the change from baseline levels (time 0) at 4 and 10 days from the initiation of anti-CDI treatment.
  Toxin kinetics (TcdA alone, TcdB alone, TcdA+TcdB) will be correlated with the duration of diarrhea. A multivariate logistic regression model will be used. The odds ratio (OR) and 95% confidence interval (CI) will be calculated. The Spearman correlation coefficients and Wilcoxon rank sum tests will be used to determine whether TcdA and TcdB levels could be associated with the duration of diarrhea.
Correlation between toxins levels and the recurrence rate | Determination of serum toxin kinetics will be evaluated by the change from baseline levels (time 0) at 30 days from the cessation of diarrhea.
  Toxin kinetics (TcdA alone, TcdB alone, TcdA+TcdB) will be correlated with the recurrence rate. A multivariate logistic regression model will be used to assess predictors of poor outcome of CDI. The odds ratio (OR) and 95% confidence interval (CI) will be calculated.
  The Spearman correlation coefficients and Wilcoxon rank sum tests will be used to determine whether TcdA and TcdB levels could be associated with the recurrence rate.
Correlation between toxins levels and mortality rate | Time-to-Event measure: toxin levels versus mortality rate, from date of patient enrollment to the date of death from any cause assessed up to 12 months.
  Survival curves comparing the mortality with toxin(s) levels will be calculated using the Kaplan-Meier method and tested for significance using the log-rank test. P<0.05 will be considered statistically significant.